CLINICAL TRIAL: NCT02903342
Title: Fever and Febrile Support for Parents and Carers of Children 2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Maria Kelly, Research Pharmacist, University College Cork
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Fever1
Record Dates: First submitted 2016-08-30; First posted 2016-09-16 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Fever; Febrile Illness
Keywords: Fever; Febrile illness; Children
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Parents will be asked to read a leaflet. They will then complete a survey and re-complete the survey via telephone two weeks later.
  Interventions: Other: Leaflet
- Control (No Intervention): Parents will be asked to complete a survey and re-complete the survey via telephone two weeks later.

INTERVENTIONS:
Other: Leaflet — A leaflet designed from data obtained from previous qualitative and quantitative studies.
  Arms: Intervention

SUMMARY:
To assess the suitability and user-friendliness of an information leaflet for parents on management of fever and febrile illness in children. The purpose of the leaflet is to provide evidence-based information for parents regarding fever and febrile illness in children.

DETAILED DESCRIPTION:
The aim of this study is to assess the suitability and user-friendliness of an information leaflet for parents on management of fever and febrile illness in children. The purpose of the leaflet is to provide evidence-based information for parents regarding fever and febrile illness in children. The potential benefit of the leaflet is empowerment parents to take responsibility for monitoring their child's illness, thereby enabling parents to take effective and informed action when required.

The investigators hypothesise that provision of a user friendly information leaflet for parents increases knowledge and provides decision support to guide parents fever management.

This study will investigate the ability of an information leaflet to increase parental knowledge regarding the management of fever and febrile illness in children. Three leaflets were designed. Stakeholders were consulted to select the most appropriate leaflet prior to the beginning of the trial. One leaflet will be used in the trial.

A prospective, multi-centre, randomized, two-parallel arm, controlled trial with blinded outcome ascertainment will be conducted. Three information leaflets were designed based on a previous survey with parents in Ireland. One leaflet was selected for use as the intervention following consultation with stakeholders.

The Primary Objective of the project is to quantify if reading and understanding a leaflet on fever and febrile illness management increases parental knowledge on the subject.

ELIGIBILITY:
Inclusion Criteria:

* Parents with at least one child aged five years of age or younger at the time of recruitment.
* Parents of healthy children.

Exclusion Criteria:

* Parents who did not have at least one child aged five years of age or younger at the time of recruitment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Increase in parental knowledge regarding temperature definition for fever | 2 weeks
  Increases in correct parental definition of fever temperature detected using a questionnaire

SECONDARY OUTCOMES:
Increase in parental knowledge regarding management of fever | 2 weeks
  Increases in correct parental management of fever detected using a questionnaire
Decrease in parents alternating between antipyretics | 2 weeks
  Decreases in parents alternating between antipyretics to manage fever detected using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kelly, MPharm, MiM, Study Director — University College Cork

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelly M, Sahm L, McCarthy S, O'Sullivan R, Mc Gillicuddy A, Shiely F. Randomised controlled trial of an intervention to improve parental knowledge and management practices of fever. BMC Pediatr. 2019 Nov 19;19(1):447. doi: 10.1186/s12887-019-1808-9. PMID 31739785